CLINICAL TRIAL: NCT02652039
Title: Interactionality of State-Trait Music Preference, Individual Variability, and Music Characteristics as a Multi-Axis Paradigm for Context-Specific Pain Perception and Management
Brief Title: Interactionality of Music Preference and Individual Variables in Pain Perception and Management
Status: Completed | Type: Observational
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Xueli Tan, Presidential Graduate Research Fellow, University of Iowa
Other Study IDs: STMP - 03
Record Dates: First submitted 2016-01-06; First posted 2016-01-11 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- cancer patients
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Questionnaires

SUMMARY:
The purposes of this study were 1) to delineate any differences in general musical taste (trait) and context-specific music preference (state), as well as preferred music characteristics in cancer patients, 2) to investigate the contributions of individual variabilities, personality, behavioral coping styles, and pain levels in predicting changes from trait to state preferences and preferred music characteristics under various pain conditions.

Cancer patients were recruited to fill in questionnaires pertaining to their demographic information (age, gender, religious preference, ethnicity, music background and experience), personality traits, music preferences, preferences for music characteristics, coping styles, and pain experiences.

ELIGIBILITY:
Inclusion Criteria:

1. Stage IV cancer diagnosis
2. Between 40 - 70 years old
3. Normal or corrected hearing
4. Able to communicate (speak, comprehend, read, write) in English
5. Signed informed consent form

Exclusion Criteria:

1. Under 40 or over 70 years old
2. Not able to communicate in English
3. Uncorrected hearing loss/impairment
4. Dementia, psychosis (hallucinations, delusions) that interferes with cognitive processing (verbal and music)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Pain on the McGill Pain Questionnaire | one year

CONTACTS AND LOCATIONS:
Overall Officials: Kate Gfeller, PhD, MT-BC, Study Chair — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States